CLINICAL TRIAL: NCT05963373
Title: Pattern of Chronic Diseases in Adults Above 18years Old
Brief Title: Pattern of Chronic Disease in Adult attendantsabove18years Old in New Vally Elkharga Family Medicine Clinic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nesma Awad Khaled, Clinical professor, Assiut University
Other Study IDs: POCDIA
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Wasting Disease of Elk and Deer; Injury; Knee, Meniscus, Old Injury or Tear
MeSH Terms: conditions — Wounds and Injuries; Lacerations | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic diseased attendants above 18years old
  Interventions: Diagnostic Test: Urine analysis
- Healthy attendants
  Interventions: Diagnostic Test: Urine analysis

INTERVENTIONS:
Diagnostic Test: Urine analysis — Diagnostic test

SUMMARY:
Globally one in three of all adult suffer from multible Chronic condition six in ten adult has achronic disease and four in ten adult have twoor more.It has been calculated that 58million death in2005 approximately 35million will be aresult of chronic disease health damaging behavior tobbaco use, poor physical activity and poor eating habbits are major contributors to the leading chronic diseases the leading chronic diseases in developed countries including arthritis, cardiovascular diseases,heart attacks,stroke,cancer, diabetes,breast&colonic cancer , Aging increasing the risk of chronic diseases like dementia ,heart diseases,cancer these are the nation's leadingdrivers of illness,disability,death and health care costs.

DETAILED DESCRIPTION:
In2008 more than1,2million people died from non communicable diseases accounting for nearly 60% of all death inthe region with wide several outbreaks of hospital acquired infection in the midlle east have occurredwith substantial morbidity and mortality.Egypt currently has the third highest prevelance of obesity inMena region after saudi arabia and Emirates similar to the Hispanic and native.American population central adiposity is particularly common among egyptienand is probably inherited the Egyptian national survey individual have central obesity.this be found strongly associated with increase risk of dm and cardiovascular diseases

ELIGIBILITY:
Inclusion Criteria:

* Attendands above18years

Exclusion Criteria:

* Attendants below18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic diseased attendands
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2023-07-23 (Estimated); Primary Completion 2023-12-23 (Estimated); Study Completion 2024-06-23 (Estimated)

PRIMARY OUTCOMES:
morbidities | 6 months
  morbidities among adults above 18 years old

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Galal Mahran, Principal Investigator — Assiut University